CLINICAL TRIAL: NCT06110026
Title: Comparative Effects of Brunkow Program and Lumbar Stabilization Exercises on Pain, Range of Motion and Disability in Chronic Nonspecific Low Back Pain
Brief Title: Bronkow Program and Lumbar Stabilization Exercises in Chronic Non Specific Low Back Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/23/0146
Record Dates: First submitted 2023-10-25; First posted 2023-10-31 (Actual); Last update posted 2023-10-31 (Actual); Status verified 2023-10

CONDITIONS: Chronic Low-back Pain; Non Specific Low Back Pain
Keywords: Brunkow exercise; Disability; non-specific low back pain; pain; range of motion
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Brunkow exercise program (Experimental): Brunkow program includes Push up and stabilization against the wrists and heels,brunkow- from plank to a standing position ,plank from lying on the stomach to a sitting in a tilted position, Turning from the back to the position on all four
  Interventions: Other: Brunkow Exercise Program
- Lumbar stabilization exercises (Experimental): lumbar stabilization exercises protocol includes Diaphragmatic breathing and abdominal bracing, bridging, side plank on knees, bird dog
  Interventions: Other: Lumbar Stabilization Exercises

INTERVENTIONS:
Other: Brunkow Exercise Program — The brunkow exercise program will be comprised of four exercise programs. Each exercise will be performed with two sets of 15 reps, 10 sec per rep 40 min per day, thrice per week for a total of four weeks.
  Arms: Brunkow exercise program
Other: Lumbar Stabilization Exercises — The lumbar stabilization exercises will be comprised of four exercise programs. Each exercise will be performed with two sets of 15 reps, 10 sec per rep 40 min per day, thrice per week for a total of four weeks.
  Arms: Lumbar stabilization exercises

SUMMARY:
The aim of this study is to compare the effects of brunkow exercise program and lumbar stabilization exercises on pain, range of motion and disability in patients with chronic non- specific low back pain

DETAILED DESCRIPTION:
The majority of research studies have primarily focused on lumbar stabilization exercises used as a standard treatment with mobilization. To the best of our knowledge it has shown that lumbar stabilization exercises alone are less efficient than lumbar stabilization exercises in strengthening muscular strength and decreasing pain in female patients with persistent low back pain than lumbar stabilization exercises combined with pain neuroscience education. However, more extensive research on a range of educational and activity programs was required. Stabilization exercises with other modalities, manual techniques, mobilizations, or exercise therapy have been practiced in the treatment of chronic non specific low back pain were found effective individually, but there was a lack of comprehensive studies including randomized clinical trials directly comparing the brunkow exercises program with stabilization exercises in patients with chronic non- specific low back pain.

This study investigates and adds up an effective and evolutionary treatment protocol in the world of physical therapy for the management of chronic non-specific low back pain rather than other conventional therapy providing to the patients with chronic low back pain now a days.

ELIGIBILITY:
Inclusion Criteria:

* Age 20 to 45 years
* Both male and female
* Low back pain > 6 months
* NPRS>3
* The symptoms of pain are lessened or disappeared after bed rest, while pain symptoms are aggravated after bending over, sitting for a long time, or standing for a long time.

Exclusion Criteria:

* Pelvic bone fracture
* Pregnancy
* Pelvic implants
* Lumbosacral disc herniation
* Sacroiliac joint inflammation
* Lumbar spine fracture
* Inflammatory bowel disease
* Malignancy
* Ankylosing spondylitis

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2023-05-08 (Actual); Primary Completion 2023-12-23 (Estimated); Study Completion 2024-01-08 (Estimated)

PRIMARY OUTCOMES:
Numeric rating scale (NRS-11) | 4 weeks
  It is is an eleven-point scale in which the end points are the extremes of no pain at all (score of 0) and the worst pain the patient has ever experienced (score of 10). NRS-11 pain severity score of "4" is frequently given special significance in this regard, suggesting it as a potential threshold value for pain severity in clinical practice. (28).
  This scale has high reliability (0.95-0.96) and validity (0.86-0.96).
Modified oswestry disability index | 4 weeks
  The ODI is a disease-specific disability measure is used to establish a level of disability, stage a patient's acuity status and monitor change over time. The ODI is made up of 10 questions. Each question is scored from 0-5 (minimum to maximum). This tool is considered as a gold standard for back pain functional. Test-retest reliability has been shown to be high. Values range from r= 0.83 to 0.99 and vary according to the time interval between measurements. ODI = (Sum of items scored/Sum of sections answered) X 100
Inclinometer | 4 weeks
  Inclinometers are portable, lightweight, and inexpensive pieces of equipment that are used to measure range of motion, like goniometry.1 Inclinometers are typically found in clinics and are used as a part of a physical examination. An intraclass correlation coefficient (ICC) was found to be between 0.87- 0.95. Range of motion is the measurement of movement around a specific joint or body part.

CONTACTS AND LOCATIONS:
Overall Officials: Humera Mubashar, MSPT, Principal Investigator — Riphah International University
Locations (1):
- University of Lahore Teaching Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Orrock PJ, Myers SP. Osteopathic intervention in chronic non-specific low back pain: a systematic review. BMC Musculoskelet Disord. 2013 Apr 9;14:129. doi: 10.1186/1471-2474-14-129. PMID 23570655
- [Background] Savigny P, Watson P, Underwood M; Guideline Development Group. Early management of persistent non-specific low back pain: summary of NICE guidance. BMJ. 2009 Jun 4;338:b1805. doi: 10.1136/bmj.b1805. No abstract available. PMID 19502217
- [Background] Garcia JB, Hernandez-Castro JJ, Nunez RG, Pazos MA, Aguirre JO, Jreige A, Delgado W, Serpentegui M, Berenguel M, Cantemir C. Prevalence of low back pain in Latin America: a systematic literature review. Pain Physician. 2014 Sep-Oct;17(5):379-91. PMID 25247896
- [Background] Nijs J, Apeldoorn A, Hallegraeff H, Clark J, Smeets R, Malfliet A, Girbes EL, De Kooning M, Ickmans K. Low back pain: guidelines for the clinical classification of predominant neuropathic, nociceptive, or central sensitization pain. Pain Physician. 2015 May-Jun;18(3):E333-46. PMID 26000680
- [Background] Forster M, Mahn F, Gockel U, Brosz M, Freynhagen R, Tolle TR, Baron R. Axial low back pain: one painful area--many perceptions and mechanisms. PLoS One. 2013 Jul 2;8(7):e68273. doi: 10.1371/journal.pone.0068273. Print 2013. PMID 23844179
- [Background] Violante FS, Mattioli S, Bonfiglioli R. Low-back pain. Handb Clin Neurol. 2015;131:397-410. doi: 10.1016/B978-0-444-62627-1.00020-2. PMID 26563799
- [Background] Waseem M, Karimi H, Gilani SA, Hassan D. Treatment of disability associated with chronic non-specific low back pain using core stabilization exercises in Pakistani population. J Back Musculoskelet Rehabil. 2019;32(1):149-154. doi: 10.3233/BMR-171114. PMID 30248035
- [Background] Faas A. Exercises: which ones are worth trying, for which patients, and when? Spine (Phila Pa 1976). 1996 Dec 15;21(24):2874-8; discussion 2878-9. doi: 10.1097/00007632-199612150-00016. PMID 9112711
- [Background] Mujic Skikic E, Trebinjac S, Sakota S, Avdic D. The effects of McKenzie and Brunkow exercise program on spinal mobility comparative study. Bosn J Basic Med Sci. 2004 Feb;4(1):62-8. doi: 10.17305/bjbms.2004.3466. PMID 15628984
- [Background] Yeom S, Jeong H, Lee H, Jeon K. Effects of Lumbar Stabilization Exercises on Isokinetic Strength and Muscle Tension in Sedentary Men. Bioengineering (Basel). 2023 Mar 8;10(3):342. doi: 10.3390/bioengineering10030342. PMID 36978733
- [Background] Skikic EM, Trebinjac S, Sakota S, Avdic D, Delic A. Brunkow exercises and low back pain. Bosn J Basic Med Sci. 2004 Oct;4(4):37-41. doi: 10.17305/bjbms.2004.3359. PMID 15628994
- [Background] Lee HS, Kim DJ, Oh Y, Min K, Ryu JS. The effect of individualized gradable stabilization exercises in patients with chronic low back pain: Case-control study. J Back Musculoskelet Rehabil. 2016 Jun 17;29(3):603-10. doi: 10.3233/BMR-160724. PMID 27341643
- [Background] Kim CR, Park DK, Lee ST, Ryu JS. Electromyographic Changes in Trunk Muscles During Graded Lumbar Stabilization Exercises. PM R. 2016 Oct;8(10):979-989. doi: 10.1016/j.pmrj.2016.05.017. Epub 2016 Jun 16. PMID 27317910
- [Background] Lee K. Motion Analysis of Core Stabilization Exercise in Women: Kinematics and Electromyographic Analysis. Sports (Basel). 2023 Mar 10;11(3):66. doi: 10.3390/sports11030066. PMID 36976952
- [Background] Kim KS, An J, Kim JO, Lee MY, Lee BH. Effects of Pain Neuroscience Education Combined with Lumbar Stabilization Exercise on Strength and Pain in Patients with Chronic Low Back Pain: Randomized Controlled Trial. J Pers Med. 2022 Feb 17;12(2):303. doi: 10.3390/jpm12020303. PMID 35207790
- [Background] Gianola S, Bargeri S, Del Castillo G, Corbetta D, Turolla A, Andreano A, Moja L, Castellini G. Effectiveness of treatments for acute and subacute mechanical non-specific low back pain: a systematic review with network meta-analysis. Br J Sports Med. 2022 Jan;56(1):41-50. doi: 10.1136/bjsports-2020-103596. Epub 2021 Apr 13. PMID 33849907
- [Background] Akodu AK, Nwanne CA, Fapojuwo OA. Efficacy of neck stabilization and Pilates exercises on pain, sleep disturbance and kinesiophobia in patients with non-specific chronic neck pain: A randomized controlled trial. J Bodyw Mov Ther. 2021 Apr;26:411-419. doi: 10.1016/j.jbmt.2020.09.008. Epub 2020 Oct 3. PMID 33992276
- [Background] Alhakami AM, Davis S, Qasheesh M, Shaphe A, Chahal A. Effects of McKenzie and stabilization exercises in reducing pain intensity and functional disability in individuals with nonspecific chronic low back pain: a systematic review. J Phys Ther Sci. 2019 Jul;31(7):590-597. doi: 10.1589/jpts.31.590. Epub 2019 Jul 9. PMID 31417227
- [Background] 20. Pysna J, Pysny L, Petru D, Cihlar D, editors. PHYSIOTHERAPEUTICAL METHODS IN THE PREVENTION OF FUNCTIONAL DISORDERS OF THE MUSCULOSKELETAL SYSTEM-A NEW TREND IN TEACHING REMEDIAL PHYSICAL EDUCATION TO UNIVERSITY STUDENTS. ICERI2019 Proceedings; 2019: IATED.
- [Background] Gomes-Neto M, Lopes JM, Conceicao CS, Araujo A, Brasileiro A, Sousa C, Carvalho VO, Arcanjo FL. Stabilization exercise compared to general exercises or manual therapy for the management of low back pain: A systematic review and meta-analysis. Phys Ther Sport. 2017 Jan;23:136-142. doi: 10.1016/j.ptsp.2016.08.004. Epub 2016 Aug 18. PMID 27707631
- [Background] Bhadauria EA, Gurudut P. Comparative effectiveness of lumbar stabilization, dynamic strengthening, and Pilates on chronic low back pain: randomized clinical trial. J Exerc Rehabil. 2017 Aug 29;13(4):477-485. doi: 10.12965/jer.1734972.486. eCollection 2017 Aug. PMID 29114516
- [Background] 23. Nasreen A, Majeed Z, Awan MAH, Maqbool S, Asghar HMU, Tahir H, et al. Comparison Of The Effectiveness Of Back School Exercises And Mckenzie Exercises In The Treatment Of Chronic Low Back Pain; A Randomized Controlled Trial" RCT: Back School Exercises and Mckenzie Exercises in The Treatment of Chronic Low Back Pain. Pakistan BioMedical Journal. 2022:112-6.
- [Background] Chiarotto A, Koes BW. Nonspecific Low Back Pain. N Engl J Med. 2022 May 5;386(18):1732-1740. doi: 10.1056/NEJMcp2032396. No abstract available. PMID 35507483
- [Background] Zhou X, Yang J, Ma QY, Guo Y, He KJ, Shen LB, Fan Q, Philip CKC, Keng TB, Celia TIC, Bauer BA, Chen JX. The effectiveness of Tuina in managing chronic non-specific low back pain: A protocol of a multicenter international randomized controlled trial. Medicine (Baltimore). 2022 Feb 18;101(7):e28883. doi: 10.1097/MD.0000000000028883. PMID 35363203
- [Background] Ahmed UA, Maharaj SS, Van Oosterwijck J. Effects of dynamic stabilization exercises and muscle energy technique on selected biopsychosocial outcomes for patients with chronic non-specific low back pain: a double-blind randomized controlled trial. Scand J Pain. 2021 Feb 24;21(3):495-511. doi: 10.1515/sjpain-2020-0133. Print 2021 Jul 27. PMID 33641272
- [Background] 27. Kahl C, Cleland JA. Visual analogue scale, numeric pain rating scale and the McGill pain Questionnaire: an overview of psychometric properties. Physical therapy reviews. 2005;10(2):123-8.
- [Background] Al-Hadidi F, Bsisu I, AlRyalat SA, Al-Zu'bi B, Bsisu R, Hamdan M, Kanaan T, Yasin M, Samarah O. Association between mobile phone use and neck pain in university students: A cross-sectional study using numeric rating scale for evaluation of neck pain. PLoS One. 2019 May 20;14(5):e0217231. doi: 10.1371/journal.pone.0217231. eCollection 2019. PMID 31107910
- [Background] 29. Waqar S, Khalid M, Khalid N. EFFECTIVENESS OF ELONGATION LONGITUDINAUX AVEC DECOAPTION OSTEOARTICULAIRE IN CORRECTING FORWARD HEAD POSTURE: soi: 21-2017/re-trjvol06iss01p284. The Rehabilitation Journal. 2022;6(01):284-9.
- [Background] Vianin M. Psychometric properties and clinical usefulness of the Oswestry Disability Index. J Chiropr Med. 2008 Dec;7(4):161-3. doi: 10.1016/j.jcm.2008.07.001. PMID 19646379
- [Background] Kolber MJ, Pizzini M, Robinson A, Yanez D, Hanney WJ. The reliability and concurrent validity of measurements used to quantify lumbar spine mobility: an analysis of an iphone(R) application and gravity based inclinometry. Int J Sports Phys Ther. 2013 Apr;8(2):129-37. PMID 23593551